CLINICAL TRIAL: NCT06239207
Title: Efficacy and Safety of Exosomes Versus Platelet Rich Plasma in Patients of Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr Alina Abbass, Senior Registrar Dermatology, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2023/1181/SIMS
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Androgenetic Alopecia
Keywords: Exosomes, Platelet Rich Plasma, Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study in which two or more groups of participants receive different interventions. Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial. Assignment to a group usually is randomized. Study participants are only exposed to the treatment that is assigned to the particular study arm they are enrolled in. So in this study the patients are randomized into two groups by paper lottery method. After regional nerve block under aseptic conditions, Group A patients are injected exosomes intradermally at a strength of 2 to 10 billion particles/5ml, at a dose of 0.1 ml/cm2 of scalp, and group B patients are injected PRP intradermally in scalp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosomes (Experimental): Group A patients are injected exosomes 2 session 3 months apart, intradermally at a dose of 0.1 ml/cm2 of scalp. Exosomes used are GFC CELL(TM) EXO SCALP KIT
  Interventions: Biological: Exosomes GFC CELL EXO SCALP KIT (Leuco Exo 97%)
- B PRP (Active Comparator): PRP 4 sessions 1 months apart. Group B patients are injected PRP intradermally in scalp. Uunder aseptic around 10ml of blood is collected from the median cubital vein and is transferred into a sodium citrate tube. Then the tubes are rotated in a centrifuge machine at 1500 RPM for 10 minutes.It separates the blood into 2 layers: the lower RBC layer; the upper plasma layer buffy coat. The buffy coat was transferred into another test tube. This tube was again subjected to a second centrifugation at 4000 RPM for 10 minutes. Both the upper layer containing platelet poor plasma and the lower layer of the PRP was collected. The plasma is filled into insulin syringe and then injected evenly into the affected areas of the scalp. Multiple PRP injections of 0.1 mL were given at each site in a linear pattern 1 cm apart
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Exosomes GFC CELL EXO SCALP KIT (Leuco Exo 97%) — Exosomes used are GFC CELL, consist of Leuco exo 97% having GFC CELL EXO SCALP 9700 powder and EXO SCALP Pep9 solution
  Arms: Exosomes
Biological: Platelet Rich Plasma — PRP is prepared under aseptic precautions, around 10ml of blood is collected in PRP tubes which are rotated in a centrifuge machine at 1500 RPM for 10 minutes. Which separates the blood into 2 layers: the lower RBC layer; the upper acellular plasma layer. The buffy coat along with the plasma was collected with a pipette and transferred into another test tube underwent 2nd spin at 4000 RPM for 10 min. This PRP was collected in another clean tube to be used as plasma
  Arms: B PRP

SUMMARY:
Androgenetic alopecia is a common condition affects both genders. Patients of androgenetic alopecia following inclusion criteria will be enrolled after ethical approval and informed consent. Pre-treatment assessment will be done by Physian Global assessment, Patient global assessment and hair density by trichoscopy of areas under treatment. Patients will be categorized in 2 groups. Group A receiving exosomes 1session intradermally in scalp after nerve block and group B receiving PRP 2 sessions of PRP 1 month apart intradermally in scalp after nerve block. Patients will receive exosomes at strength of 2 to 10 billion particles/5ml with 0.1 ml/cm2. Follow up will be done after 1 month, 2 months, 3 months, 5 months and 6 months of completion of treatment to assess hair growth and reduce hair fall by Physian Global assessment (PGA), Patient global assessment (PtGA) and trichography. Clinical response will be graded as satisfactory (< 25%), good (25-50%) or excellent (> 50%) improvement. Details will be entered on predesigned proforma. Data will be entered and analyzed using SPSS 27. Means will be calculated for quantitative variables, frequencies for qualitative variables like pre- and post treatment response. Data will be stratified for role of effect modifiers

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is a common condition that affects up to 50 percent of males and females. It is characterized by progressive loss of terminal hair of the scalp any time after puberty. It has a very typical distribution in both males and females. In males, hair loss is mostly on vertex and frontotemporal regions, while in women the frontal hairline is mostly involved with diffuse hair loss at the crown and top of head. Currently, FDA approved treatments are topical minoxidil and oral finasteride. But due to its adverse effects, most patients refuse to take this drug. Platelet rich plasma (PRP) is currently effective alternate therapy used very commonly. PRP is autologous concentration of platelets, having multiple growth factors in their alpha granules, injected intradermally in scalp. There is another emerging treatment modality which is exosomes. Exosomes are 30-150nm extracellular vesicles (EVs) derived from various mesenchymal stem cells (MSCs). Exosomes contain various proteins, nucleic acids and various cell mediators and growth factors. They have same biological properties as that of their parent derived cell along with advantages of small size, easy penetration of biological membranes, low immunogenicity, easy storage, and no tumorization. Recently, exosomes have been genetically modified so that they can exhibit better therapeutic properties, such as enriched active ingredients, targeted delivery, and physiological barrier to penetration. Because of their properties they have roll in hair growth. Exosomes are providing promising results in patients of androgenetic alopecia. Both PRP and exosome therapy has found to be effective in various studies across the globe. Very less literature is found on comparison of these two treatment modalities specially in the world.

Learning Objective is to compare the efficacy and safety of PRP and Exosomes in patients of Androgenetic alopecia.

It is a randomized clinical trial going on in Dermatology department of Services hospital Lahore, Pakistan. After getting approval from Ethical Review Board.

Pre-treatment assessment is done by hair pull test, global physician assessment, patient global assessment and hair density by trichoscopy of the involved areas of scalp. The patients are randomized into two groups by paper lottery method. After regional nerve block under aseptic conditions, Group A patients are injected exosomes intradermally at a strength of 2 to 10 billion particles/5ml, at a dose of 0.1 ml/cm2 of scalp, and group B patients are injected PRP intradermally in scalp. Exosomes used are GFCCELLTM EXO SCALP KIT. PRP is prepared under aseptic precautions, around 10ml of blood is collected from the median cubital vein and is transferred into a sodium citrate tube. Then the tubes are rotated in a centrifuge machine at 1500 RPM for 10 minutes. This first centrifugation is called "soft spin," which separates the blood into 2 layers: the lower RBC layer; the upper acellular plasma layer which is further subdivided into an upper layer which contains platelet poor plasma and a lower layer which contains platelet rich plasma also known as the buffy coat. The buffy coat along with the plasma was collected with a pipette and transferred into another test tube. This tube was again subjected to a second centrifugation at 4000 RPM for 10 minutes, called "hard spin." This allows the platelets to settle at the bottom of the tube. Both the upper layer containing platelet poor plasma and the lower layer of the PRP was collected in another clean tube. The plasma is filled into insulin syringe and then injected evenly into the affected areas of the scalp. Multiple PRP injections of 0.1 mL were given at each site in a linear pattern 1 cm apart. The patients are followed monthly after the first treatment session for 6 months. The primary efficacy endpoints of this study are increse in hair regrowth assessed by Global physician assessment and patient global assessment on scale of three ( <25% as satisfactory, 25-50% as good response, >50% as excellent response) and number of hairs which are calculated by trichoscopy. Demographic data and pretreatment parameters are recorded on a predesigned proforma. Data is entered and analyzed using SPSS vs 20.

ELIGIBILITY:
Inclusion Criteria:

* All patients with androgenetic alopecia
* age from 18 to 70 years
* Sex: male and female

Exclusion criteria:

* Patient with platelets disorders, thrombocytopenia
* Patients using anti-platelet therapy
* Use of pharmacological therapeutics targeting AGA as Finasteride®, use of topical medicines as lotions as Minoxidil®, retinoid, or corticosteroids in the earlier year.
* Patients with bone marrow aplasia, uncontrolled diabetes, sepsis, cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
More than 25% increase in hair density | 6 months after last session
  hairs per cm square measured by trichoscopy

SECONDARY OUTCOMES:
> 25% improvement response in Physician Global assesment | 6 months after last sessions
  3 points scoring system, score 1 satisfactory response <25% improvement, score 2 25-50% improvement good response, score 3 >50% improvement excellent response
> 25% improvement response in Patient Global assesment | 6 months after last sessions
  3 points scoring system, score 1 satisfactory response <25% improvement, score 2 25-50% improvement good response, score 3 >50% improvement excellent response

CONTACTS AND LOCATIONS:
Overall Officials: Alina Abbass, MBBS, FCPS, Principal Investigator — Services Institute of medical Sciences
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No